CLINICAL TRIAL: NCT01481857
Title: Influence of Thoracolumbar Proprioceptive Support in the Segmental Stabilization Training
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Universidade Federal do Piauí (Other)
Responsible Party: Principal Investigator, Fuad Ahmad Hazime, Assistant Professor at School of Physiotherapy, Universidade Federal do Piauí
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0378.0.045.000-10
Record Dates: First submitted 2011-11-23; First posted 2011-11-30 (Estimated); Last update posted 2011-11-30 (Estimated); Status verified 2011-11

CONDITIONS: Transversus Abdominis Activation
MeSH Terms: interventions — Proprioception

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Thoracolumbar proprioception (Experimental)
  Interventions: Other: Segmental trunk exercise associated with proprioception
- Segmental Stabilization (Experimental)
  Interventions: Other: Segmental trunk exercise

INTERVENTIONS:
Other: Segmental trunk exercise associated with proprioception — Proprioceptive exercise
  Arms: Thoracolumbar proprioception
Other: Segmental trunk exercise — Segmental trunk exercise
  Arms: Segmental Stabilization

SUMMARY:
Proprioceptive training has been shown to be effective in increasing the efficiency of motor-sensory tissues that stabilize the trunk. The investigators hypothesis is that proprioceptive support do influence in the activation of the transversus abdominis muscle (TrA) during segmental stabilization training.

ELIGIBILITY:
Inclusion Criteria:

* healthy subjects

Exclusion Criteria:

* subjects with any kind of disease

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2011-02; Primary Completion 2011-03 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Activation of transversus abdominis | Two Weeks
  Activation of transverus abdominis will be assessed by the biofeedback pressure unit.Pressure biofeedback units consist of a combined inflation bulb connected to a pressure cell.

CONTACTS AND LOCATIONS:
Locations (1):
- Fuad Ahmad Hazime, Parnaíba, Piauí, Brazil